CLINICAL TRIAL: NCT04550000
Title: A Multi-center Sample Collection Study in Patients With Suspected Melanoma Utilizing DermTech's Non-invasive Adhesive Patch Biopsy Kits
Brief Title: Sample Collection Study in Patients With Suspected Melanoma Utilizing DermTech's Non-invasive Adhesive Patch Biopsy Kits
Status: Completed | Type: Observational
Sponsor: DermTech (Other)
Responsible Party: Sponsor
Other Study IDs: 19-01
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2021-03

CONDITIONS: Melanoma (Skin); Pigmented Skin; Nevus
Keywords: Pigmented Lesion Assay (PLA); DermTech
MeSH Terms: conditions — Melanoma; Pigmentation Disorders; Nevus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin issue collected non-invasively will the extracted and nucleic acids isolated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multi-center sample collection study in patients presenting with pigmented lesion(s) suspicious for melanoma. All suspicious lesions should meet at least one of the "ABCDE" criteria.

DETAILED DESCRIPTION:
A multi-center sample collection study in patients presenting with pigmented lesion(s) suspicious for melanoma. All suspicious lesions should meet at least one of the "ABCDE" (asymmetry, border, color, diameter, evolving) criteria. Patients will be consented for the study and screened against the inclusion and exclusion criteria. Once the patient is determined to be acceptable for the study they will be assigned a unique patient number and tissue collection will begin. Tissue from the lesion will be collected using DermTech's non-invasive adhesive patch kit according to the instructions for use followed by surgical biopsy. Digital dermoscopy of the lesion is preferred but not required.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 21 years of age
2. Have a pigmented lesion suspicious for melanoma the pigmented lesion meets at least one of the "ABCDE" criteria
3. The pigmented lesion mst be at least 3mm and not more than 16mm in diameter
4. Patient is willing to follow the start of care to test and treat the pigmented lesion as determined by the treating physician
5. Willing to have DermTech adhesive patch biopsies performed
6. Must be able to complete study procedures as required by the protocol
7. Willing to provide informed consent to participate in this trial

Exclusion Criteria:

1. Require a surgical biopsy or excision of the lesion of interest prior to the DermTech non-invasive patch biopsy(ies)
2. Has an ulcerated or bleeding lesion that could confound the biopsy results
3. Has a suspicious lesion(s) in an area that was previously surgically biopsied
4. Has a lesion that is classified as "clinically" evident melanoma appropriate for excision
5. The lesion to be sampled is on the mucosal surface, palmoplantar surface or other area where adhesive patch biopsies cannot be performed
6. Has a known sensitivity to adhesive patches
7. Any significant medical condition that would indicate an unreasonable risk to the patient or potential interference with the study
8. Lesion is in a location were sufficient removal of non-vellus hair cannot be achieved (e.g., scalp)
9. Suspected non-melanoma skin cancer
10. Patients with contraindication(s) to surgical biopsy -

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll all patients who present to a physician for examination of lesions suspicsion for melanoma
Sampling Method: Non-Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Up to 1000 samples will be compared for gene expression analysis results compared to biopsy findings. | Samples will be extracted and analyzed once up to 1000 samples have been collected and compared to surgical biopsy reports. Analysis results are expected in 2021
  gene expression associated with melanoma vs non-melanoma compared to surgical biopsy
Up to 1000 samples will be compared to biopsy results for DNA mutations | Samples will be extracted and analyzed once up to 1000 samples have been collected and compared to surgical reports and DNA mutation analysis. Analysis results are expected in 2021
  Dna mutations associated with more aggressive forms of melanoma

CONTACTS AND LOCATIONS:
Overall Officials: James Rock, Study Director — DermTech
Locations (2):
- United States (2):
  - Dermatologic Surgery Center, Chevy Chase, Maryland
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Result] Yao Z, Allen T, Oakley M, Samons C, Garrison D, Jansen B. Analytical Characteristics of a Noninvasive Gene Expression Assay for Pigmented Skin Lesions. Assay Drug Dev Technol. 2016 Aug;14(6):355-63. doi: 10.1089/adt.2016.724. PMID 27505074
- [Result] Gerami P, Yao Z, Polsky D, Jansen B, Busam K, Ho J, Martini M, Ferris LK. Development and validation of a noninvasive 2-gene molecular assay for cutaneous melanoma. J Am Acad Dermatol. 2017 Jan;76(1):114-120.e2. doi: 10.1016/j.jaad.2016.07.038. Epub 2016 Oct 1. PMID 27707590